CLINICAL TRIAL: NCT01741883
Title: Clinical Application of Nocebo Research: Optimizing Expectations of Breast Cancer Patients to Prevent Nocebo Side Effects and Decrease of Quality of Life During Adjuvant Endocrine Therapy (DFG, NE 1635/2-1)
Brief Title: Side Effect Prevention Training (SEPT) for Nocebo Effects in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Philipps University Marburg (Other)
Collaborators: University of Hamburg-Eppendorf (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Yvonne Nestoriuc, PhD., Prof. Dr., Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DFG NE 1635/2-1
Record Dates: First submitted 2012-12-04; First posted 2012-12-05 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Female Breast Cancer
Keywords: Randomized Controlled Trial; Patients´ Expectations; Breast Cancer; Adjuvant Endocrine Treatment; Nocebo
MeSH Terms: conditions — Breast Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Medical Care and Information (No Intervention): Patients receive standard treatment protocol for breast cancer patients and additional oral and written information about adjuvant endocrine treatment.
- Side effect prevention training (SEPT) (Experimental): Patients receive standard medical care and a brief behavioral intervention that targets patients' response and coping expectations while starting with adjuvant endocrine treatment.
  Interventions: Behavioral: Side effect prevention training (SEPT)
- Attention Control group (ACG) (Active Comparator): Patients receive standard medical care and a comparable amount of therapist´s attention (common and unspecific factors) to the intervention group without targeting patients´ expectations.
  Interventions: Behavioral: Attention Control group (ACG)

INTERVENTIONS:
Behavioral: Side effect prevention training (SEPT) — SEPT is aimed to optimize patients' response expectations before the start of pharmacotherapy to prevent nocebo side effects during adjuvant endocrine treatment. SEPT is a three session cognitive-behavioural training. It includes psychoeducation about AET to provide a realistic view on AET, reduction of concerns about side effects and strengthening of necessity beliefs. Further contents are side effect management training and problem solving to enhance self-efficacy expectations about coping as well as imagination training to integrate positive aspects of medication into daily life.
  Arms: Side effect prevention training (SEPT)
Behavioral: Attention Control group (ACG) — Supportive therapy includes common or unspecific factors such as elicitation of affect, a treatment context, empathy, reflective listening, and feeling understood. Supportive therapy thus provides a control condition for common factors and therapist attention, while lacking the specific intervention part. It will be delivered in the same frequency and at the same time points as the side effect prevention training (three individual sessions and three booster telephone calls).
  Other Names: Supportive therapy
  Arms: Attention Control group (ACG)

SUMMARY:
The purpose of this study is to evaluate a side effect prevention training (SEPT) that optimizes patients' response expectations before the start of adjuvant endocrine treatment (AET) to prevent nocebo side effects and enhance quality of life during longer term drug intake.

DETAILED DESCRIPTION:
The majority of breast cancer patients discontinue today's standard adjuvant treatment (endocrine therapy) due to side effects and reduced quality of life. Thereby, most side effects are unspecific, thus, not related to the specific pharmacological action of the drug, but to the individual treatment context and patients´ expectations (nocebo effects). The aim of this study is to evaluate a side effect prevention training (SEPT) that optimizes patients' response expectations before the start of pharmacotherapy to prevent nocebo side effects during longer term drug intake. Using a randomized trial, we will study the time course of response expectations and side effects in breast cancer patients receiving either SEPT, standard medical care or an attention-control intervention ("supportive therapy") before the start of adjuvant endocrine therapy. We will analyze the effects of changing pre-treatment expectations on cancer-treatment related side effects, quality of life and adherence 3 and 6 months after the start of endocrine therapy. Moderator analyses will be used to determine predictors of non-specific medication side effects and patients that are at high risk of experiencing them. Furthermore, we will explore the mediating influence of coping behaviours, thereby providing insights into pathways of clinical nocebo effects. The study findings promise significant advances in the clinical application of nocebo research with strong implications for clinical and research practice.

ELIGIBILITY:
Inclusion Criteria:

* Women with estrogen receptor positive breast cancer scheduled to start first-line adjuvant endocrine therapy with Tamoxifen (+/- GnRH) or a third generation Aromatase inhibitor at the Breast Cancer Centre
* Sufficient knowledge of German language and ability to give informed consent
* Age of 18 and more

Exclusion Criteria:

* Presence of a serious comorbid psychiatric condition (schizophrenia or addiction, severe depression or anxiety)
* Presence of a life threatening comorbid medical condition

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Side Effects (General Assessment of Side Effects, GASE) | Baseline, 3 and 6 months after the start of adjuvant endocrine therapy (AET)
  Side Effects 3 and 6 months after the start of adjuvant endocrine therapy, controlled for baseline symptoms, staging, age, medication

SECONDARY OUTCOMES:
Change in Patients Expectations (General Assessment of Side Effects-Expect/Cope, Gase-Expect/Cope; Brief Illness Perceptions Questionnaire, B-IPQ; Beliefs about medicine questionnaire, BMQ-D) | Baseline and 5 weeks after surgery, before start of adjuvant endocrine therapy
  Change in patients expectations from baseline/pre-intervention (expected average 2 weeks after surgery) to post-intervention (expected average 5 weeks after surgery) and prospective expectations 3 and 6 months after the start of adjuvant endocrine therapy
Change in Anxiety and Depression (Hospital Anxiety and Depression Scale, HADS-D) | Baseline, 5 weeks after surgery, 3 months after the start of adjuvant endocrine therapy (AET) and 6 months after the start of AET
  Change in anxiety and depression from baseline to 5 weeks after surgery to 3 months after the start of AET to 6 months after the start of AET
Change in Fear of Progression (Fear of Progression Questionnaire-Short Form, FoP-Q-SF) | Baseline, 5 weeks after surgery, 3 months after the start of adjuvant endocrine therapy (AET) and 6 months after the start of AET
  Change in Fear of Progression from baseline to 5 weeks after surgery to 3 months after the start of AET to 6 months after the start of AET
Change in Adherence Intention and Adherence (Medication Adherence Report Scale, MARS-D) | Baseline, 5 weeks after surgery, 3 months after the start of adjuvant endocrine therapy (AET) and 6 months after the start of AET
  Change in Adherence Intention and Adherence from baseline to 5 weeks after surgery to 3 months after the start of AET to 6 months after the start of AET
Change in Quality of Life (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire with breast module, EORTC QLQ-C30 and QLQ-BR23) | Baseline, 3 and 6 months after the start of adjuvant endocrine therapy (AET)
  Change in Quality of Life from baseline to 3 months after the start of adjuvant endocrine therapy to 6 months after the start of adjuvant endocrine therapy
Change in Coping with Side Effects (General Assessment of Side Effects-Cope, GASE-Cope) | 3 and 6 months after the start of adjuvant endocrine therapy (AET)
  Change in coping with Side Effects from 3 months after the start of adjuvant endocrine therapy to 6 months after the start of adjuvant endocrine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Nestoriuc, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Winfried Rief, Prof. Dr., Principal Investigator — Philipps University Marburg, Department of Psychology, Division of Clinical Psychology and Psychotherapy; Ute-Susann Albert, Prof. Dr., Principal Investigator — Krankenhaus Nordwest, Department of Gynecology and Obstetrics
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] von Blanckenburg P, Schuricht F, Albert US, Rief W, Nestoriuc Y. Optimizing expectations to prevent side effects and enhance quality of life in breast cancer patients undergoing endocrine therapy: study protocol of a randomized controlled trial. BMC Cancer. 2013 Sep 18;13:426. doi: 10.1186/1471-2407-13-426. PMID 24047450
- [Derived] Heisig SR, Shedden-Mora MC, von Blanckenburg P, Rief W, Witzel I, Albert US, Nestoriuc Y. What do women with breast cancer expect from their treatment? Correlates of negative treatment expectations about endocrine therapy. Psychooncology. 2016 Dec;25(12):1485-1492. doi: 10.1002/pon.4089. Epub 2016 Feb 23. PMID 26913587
- See also: Homepage of the transregional DFG research unit FOR 1328: Expectation and conditioning as basic processes of the placebo and nocebo response: From neurobiology to clinical applications — http://www.placeboforschung.de